CLINICAL TRIAL: NCT05286255
Title: Safety and Tolerability of Allogeneic Umbilical Cord Derived Mesenchymal Stromal Cells (UC-MSCs) to Limit COVID Associated ComplicatioNs: an Open Label, Phase 1 Study in Hospitalized Patients (SAMPSON-1)
Brief Title: Mesenchymal Stromal Cells for COVID-19 and Viral Pneumonias
Acronym: SAMPSON-1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Medical University of South Carolina (Other)
Collaborators: Pandorum International, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115966
Record Dates: First submitted 2022-03-16; First posted 2022-03-18 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: COVID-19 Pneumonia; Viral Pneumonia
Keywords: Mesenchymal Stromal Cells; ARDS; COVID-19; MSC; Stem Cells
MeSH Terms: conditions — Pneumonia, Viral; COVID-19

STUDY DESIGN:
Intervention Model Description: Open label, single group, Phase 1 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Allogeneic Mesenchymal Stromal Cell infusion (Experimental): Intravenous infusion of 1.25-1.5 x 10^6 cells/kg with a maximal dose of 100 x 10^6 cells on days 1 and 3 after study enrollment.
  Interventions: Biological: Allogeneic Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Allogeneic Mesenchymal Stromal Cells — Intravenous MSCs 1.2-1.5 x 10^6 cells/kg on Days 1 and 3 after study enrollment

SUMMARY:
This is an open-label phase 1 clinical trial of allogeneic umbilical cord derived mesenchymal stromal cells (MSCs) for hospitalized individuals with COVID-19 or other viral pneumonias. Hospitalized individuals who are within 7 days of the onset of a viral pneumonia will be given 2 doses of MSCs at days 1 and 3 after consent. The safety of intravenous infusion will be tested and course of the oxygen response to treatment over 90 days will be evaluated.

DETAILED DESCRIPTION:
Study Design: This open-label phase 1 trial in 10 patients will assess the efficacy and safety of UC-MSCs given on day 1 and 3 in hospitalized patients with acute respiratory symptoms between 1 and 7 days after the onset of symptoms.

The following will be assessed in all subjects:

* Age, sex, comorbidities, date of symptoms, source of infection, type of admission, APACHE II score, SOFA score, Clinical status, vital signs including temperature, respiratory rate, oxygen saturation, oxygen requirement, CBC with neutrophil counts, lymphocyte count, CRP, chest imaging (CT or X-ray), location and status in hospital.
* Safety and efficacy: Day 0 (baseline), 3, and 5. Monitoring at 14, 21 and 28 days and monthly for 3 months will be obtained by telephone consult and chart review with serial laboratory.
* Serum or plasma antibody titer to SARS-CoV-2: Day 0, and 5 (additional days 14, 21 and 28 may be included, as available).
* SARS-CoV-2 PCR from nasopharyngeal swabs: Day 0 and 5. (additional day 14, 28 and 60 day samples may be tested if available or at any time when there is clinical suspicion for COVID-19 persistence).
* Outcome measures: O2 requirement (PaO2/FiO2 ratio or SpO2/FIo2), supplemental oxygen strategy (nasal cannula, high flow nasal cannula, noninvasive ventilation, intubation and invasive mechanical ventilation, neuromuscular blocking agent use, prone positioning, corticosteroids, ECMO), vasopressors, renal support, ICU LOS, ICU mortality, Hospital LOS, Hospital mortality, 28 day mortality.

Study Agent:

• Allogeneic UC-MSCs given intravenously at 1.2-1.5 x 106 cells/kg on day 1 and day 3 of study entry. A maximum dose of 100 x 106 cells would be given in each dose. All cellular product will be given with actively growing cells >24 hours from the time of thawing in the Center for Cellular Therapy (CCT) at MUSC. Any emerging FDA guidance will be followed.

Primary Safety Objective: Evaluate the safety of treatment with UC-MSCs in hospitalized patients with COVID-19 and respiratory symptoms.

Primary Safety Endpoint:

1. Rapid deterioration of respiratory or clinical status within 6 hours after transfusion of UC-MSCs

Secondary Safety Endpoints:

1. Cumulative incidence of serious adverse events during the study period
2. Transfer to intensive care unit (ICU)
3. Type and duration of respiratory support (and other ICU support)
4. ICU mortality and length of stay
5. Hospital mortality and length of stay
6. Ventilator-free days
7. 28 day mortality

Exploratory Efficacy Objective: Evaluate changes in oxygenation, progression, and regression of viral pneumonias

Efficacy Endpoint: Change from baseline in PaO2/FiO2 ratio at day 5 Biologic Samples will be serially collected to determine mechanisms of effect. Propensity matching of the cohort to the MUSC COVID-19 Biorepository population will provide a population for comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with COVID-19 respiratory symptoms and confirmation via COVID-19 SARS-CoV-2 RT-PCR testing.
2. Patient or their surrogate is willing and able to provide written informed consent and comply with all protocol requirements.
3. Diagnosis with Mild or Moderate Pneumonia not requiring mechanical ventilation: Patient must have at least one of the following features:

   i. Bilateral pneumonia present on chest radiograph or computed tomography ii. Partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) on arterial blood gas showing: >100mmHg and ≤ 300mmHg regardless of oxygen dose at time of testing.

   iii. Pulse oxygen saturation (SpO2) at rest ≤ 93% or any degree of hypoxia requiring supplemental oxygen
4. Patient agrees to storage of specimens for future testing.
5. Willingness to undergo mechanical ventilation for worsening

Exclusion Criteria:

1. Intubation with mechanical ventilation prior to study enrolment. High flow nasal cannula and non-invasive mechanical ventilation is allowed.
2. Pneumonia caused by bacteria, mycoplasma, chlamydia, legionella, fungi or other viruses
3. Obstructive pneumonia induced by lung cancer or other known causes
4. Significant comorbid illness likely to impact the outcome of COVID-19 including but not limited to active malignancy other than skin cancer.
5. Patients who are participating in other therapeutic clinical trials within 30 days of consent.
6. History of long-term use of immunosuppressive agents including prednisone dose >5mg daily over the 30 days prior to enrollment.
7. History of severe chronic respiratory disease and requirement for long-term oxygen therapy
8. Undergoing hemodialysis or peritoneal dialysis
9. Estimated or actual rate of creatinine clearance < 15 ml/min
10. History of moderate and severe liver disease (Child-Pugh score >12)
11. Substance abuse sufficient that the patient is unlikely to comply with testing requirements.
12. History of deep venous thrombosis, pulmonary embolism, cerebral vascular disease within the last 3 years
13. Known HIV, hepatitis virus, or syphilis infection
14. Co-Infection of tuberculosis, influenza virus, adenovirus and other respiratory infection virus
15. Moribund patient not expected to survive > 24hours
16. Allergy to diphenhydramine, or hydrocortisone
17. Any condition unsuitable for the study as determined by the investigators
18. Female subjects with positive pregnancy test, breastfeeding, or planning to become pregnant/breastfeed during the study period.
19. Receipt of experimental therapy for COVID-19 with the exception of convalescent plasma, dexamethasone or another corticosteroid, or remdesivir in an open label study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical deterioration | 6 hours
  Change in oxygen saturation or clinical symptoms

SECONDARY OUTCOMES:
Serious Adverse Events | 90 days
  Cumulative incidence of all serious adverse events
ICU transfer | 90 days
  Need for transfer to an intensive care unit
Respiratory support | 90 days
  Type and duration of respiratory support
Hospital mortality and length of stay | 90 days
  Hospital mortality and length of stay
Ventilator free days | 90 Days
  Days off of mechanical ventilation
28 day mortality | 28 days
  28 day mortality

OTHER OUTCOMES:
Change is PaO2/FiO2 ratio from baseline to day 5 | 5 days
  Change in oxygenation
Anti-SARS-CoV-2 titers | 14, 21 and 28 days
  Antibody titers to the SARS-CoV-2 virus
Nasopharyngeal swab SARS-CoV-2 RT-PCR | Day 5
  Rates, levels and duration of SARS-CoV-2 RNA in nasopharyngeal swabs using RT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Strange, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Biosamples are stored in the MUSC COVID-19 Biorepository
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Samples and Matching Participant data will be shared at the end of the study
Access Criteria: Email to strangec@musc.edu